CLINICAL TRIAL: NCT04185909
Title: A Prospective, Multicenter, Single Arm Clinical Study Evaluating the Use of the Renuvion Dermal System for Dermal Resurfacing
Brief Title: Renuvion Dermal System for Dermal Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-1909
Record Dates: First submitted 2019-12-03; First posted 2019-12-04 (Actual); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Wrinkle; Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All Subjects (Experimental): Subjects will be treated with the Renuvion Dermal System.
  Interventions: Device: Renuvion Dermal System

INTERVENTIONS:
Device: Renuvion Dermal System — The Renuvion® Dermal System consists of an electrosurgical generator unit, a handpiece with detachable standoffs, and a supply of helium gas. Radio Frequency (RF) energy is delivered to the handpiece by the electrosurgical generator unit and used to energize an electrode. When helium gas is passed over the energized electrode, a helium plasma is generated which allows for conduction of the RF energy from the electrode to the subject in the form of a precise helium plasma beam.

SUMMARY:
This is a multi-center, single arm, evaluator-blind prospective study of up to 55 study subjects who are seeking a procedure to reduce the appearance of wrinkles and rhytides.

DETAILED DESCRIPTION:
This is a multi-center, single arm, evaluator-blind prospective study of up to 55 study subjects who are seeking a procedure to reduce the appearance of wrinkles and rhytides. All study subjects will be treated with the Renuvion Dermal System.

The study population will consist of males and females, 30 years of age or older, requesting a procedure for the purpose of improving facial appearance by reducing facial wrinkles and rhytides. Those subjects who meet eligibility criteria and agree to provide written informed consent will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥30 years of age.
2. Subject is seeking improvement of facial appearance by reducing facial wrinkles and rhytides.
3. Subject with a facial wrinkle score rating of at least 4 on the FWS.
4. Subject with a Fitzpatrick Skin Scale score ≤III.
5. Subjects who are willing and able to take protocol allowed medications prescribed at investigator discretion which may include Keflex or Z-pack as an antibiotic, Acyclovir or Valtrex as an antiviral, Diflucan as an antifungal, Ativan or Valium for anxiety during treatment, Norco or Ultram for pain control during or post-procedure, Gabapentin, Tylenol with Codeine or NSAIDS for post-procedure pain control, and/or Antihistamines for itching during healing.
6. Subjects who are willing to have polycarbonate eye shields placed for study treatment.
7. Subject is willing and able to provide written informed consent.
8. Subject is willing and able to comply with protocol requirements, including obtaining study-required images/photos and assessments, post-care instructions, and returning for follow-up visits.
9. Subject is willing to maintain baseline skin care regimen during study participation with the exception when protocol specified ointments, moisturizers, and cleansers are required during healing stage (through approximately the 30-day follow-up). Sunblock is required throughout the study starting on approximately day 10.
10. Subject is willing to release rights to study Sponsor for the use of the photos, including in potential publication.
11. Subject is willing to abstain from other facial cosmetic procedures through the 6-month follow-up visit; examples include, but are not limited to, laser or chemical re-surfacing, dermabrasion, neuromodulator and/or filler injections, aesthetic facial surgery, etc.

Exclusion Criteria:

1. Subject with a Fitzpatrick Skin Scale score ≥IV.
2. Subject is pregnant or lactating.
3. Active HSV-1 or diabetes mellitus.
4. Active cut, wound, or infection on the skin of the face.
5. Subject has used, within 30 days prior to screening or plans to use during study participation, Accutane, Retinol, or any medication that can cause dermal hypersensitivity.
6. Subject has used, within 10 days prior to study treatment, aspirin or NSAIDs.
7. Subject has a history of autoimmune disease (excluding Hashimoto's thyroiditis).
8. Subject with a known bleeding disorder or who is on blood thinning medication that may be at risk for bleeding.
9. Subject has a known adverse reaction to lidocaine and/or epinephrine.
10. Subjects with active skin disease of the facial area or known connective tissue disease.
11. Subjects with known susceptibility to keloid formation or hypertrophic scarring.
12. Subjects with present cancerous or pre-cancerous lesions in the area to be treated.
13. Subject who, for any reason, suspects that they will not be able to complete the prescribed follow-up assessment(s).
14. Subject has had concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety and effectiveness of the study treatment method.
15. Subject is not willing to release rights to study Sponsor for the use of the photos, including in potential publication.
16. Subject is enrolled in another investigational (drug or device) clinical trial that can interfere with this study's assessments.
17. Subject has undergone a facelift procedure within 12 months prior to the screening visit.
18. Subject has received IPL, microneedling, or chemical peels within 3 months prior to the screening visit.
19. Subject has received microneedling with RF or any facial treatment with an energy-based device within 6 months prior to the screening visit.
20. Subject has received facial injections with BOTOX® or other toxins within 6 months prior to the screening visit.
21. Subject has received hyaluronic acid or calcium hydroxylapatite fillers within 4 months prior to the screening visit.
22. Subject who is a family member or employee of the investigator or sponsor.
23. Participation in any other investigational study within 30 days prior to consent.
24. Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Zimmerman, MD, Principal Investigator — Aesthetic Revolution Las Vegas
Locations (4):
- United States (4):
  - Michael Lin, MD, Sherman Oaks, California
  - Contemporary Plastic Surgery, Jacksonville, Florida
  - Holcomb-Kreithen Plastic Surgery and MedSpa, PLLC, Sarasota, Florida
  - Aesthetic Revolution Las Vegas, Las Vegas, Nevada

REFERENCES:
- [Derived] Holcomb JD, Doolabh V, Lin M, Zimmerman E. High energy, double pass helium plasma dermal resurfacing: A prospective, multicenter, single-arm clinical study. Lasers Surg Med. 2022 Jul;54(5):648-662. doi: 10.1002/lsm.23524. Epub 2022 Feb 16. PMID 35170772

RESULTS

PARTICIPANT FLOW:
Groups:
- Full-face Renuvion Dermal System Treatment: Perioral, Forehead, Nose, and Cheek zones were treated with two (2) passes of the plasma beam at 40% power and 4 liters/minute helium flow utilizing the appropriate standoff with one pass done horizontally and the other pass done perpendicular. The Periorbital zone was treated with one (1) or two (2) passes, based on the investigator's discretion, 20% power and 4 liters/minute helium flow utilizing the appropriate standoff (spacer) with up to 2 passes done horizontally or only in one direction. The Jawline/Mandibular Border was treated with one (1) or two (2) passes, based on the investigator's discretion, at 20% - 40% power and 4 liters/minute helium flow using the appropriate standoff and a treatment pattern in a variable motion to achieve blending. For areas that were treated with a 2nd pass, the eschar was wiped away entirely prior to start of the 2nd pass.
Period: Overall Study
Arm/Group | Full-face Renuvion Dermal System Treatment
Started | 55
Completed | 54
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Age, Customized [Mean (Standard Deviation); unit: years]
  Adults 30 yrs of age or older who signed informed consent and who met inclusion/exclusion criteria. | 64.5 (7.0)
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Adults 30 yrs of age or older who signed informed consent and who met inclusion/exclusion criteria. | 65.0 [61 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (4.0)
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 24.3 [22 to 27]
Fitzpatrick Skin Type Scale (FST) [Count of Participants; unit: Participants] — Assessment of subject's skin color was determined prior to study procedure by the investigator using the FST. The scale delineates skin color into categories.
  Type I: White skin that never tans and always burns easily Type II: White skin that tans slightly and always burns easily Type III: Light brown skin that tans gradually and can burn moderately Type IV: Moderately brown skin that tans well and burns slightly Type V: Dark brown skin that tans profusely and burns rarely Type VI: Black skin with deep pigmentation that never burns
  Participants
    Type I | 4
    Type II | 38
    Type III | 13
Fitzpatrick Wrinkle and Elastosis Scale (FWS) [Count of Participants; unit: Participants] — Assessment of each subject's wrinkles categorized into Class I-III and Scores 1-9.
  Class I: Fine wrinkles Class II: Fine to moderate depth wrinkles, Moderate number of lines Class III: Fine to deep wrinkles, numerous lines, with or without redundant skin folds.
  Score 1-3: Mild- fine texture changes with subtly accentuated skin lines. Score 4-6: Moderate- distinct papular elastosis and dyschromia. Score 7-9: Severe- Multipapular and confulent elastosis approaching or consistent with cutis rhomboidalis.
  Participants
    Class II: Score 5 | 1
    Class II: Score 6 | 14
    Class III: Score 7 | 12
    Class III: Score 8 | 19
    Class III: Score 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Independent Photo Reviewer Fitzpatrick Wrinkle and Elastosis Scale (FWS)
Description: The FWS is a clinically validated assessment tool used to assess skin wrinkle severity and elastosis on a scale from 1 through 9, where the lower the value, the better the outcome. Three Independent Photographic Reviewers were blinded to the study subject's visit (Day 90 follow-up visit) and performed photographic assessments of each subject's wrinkle depth in the treated zones.
Time Frame: 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants | 55
Statistical Analysis 1: Comparison: Full-face Renuvion Dermal System Treatment; Test type: Superiority; p < .0001, Fisher Exact

2. Other Pre Specified Outcome: Independent Photographic Reviewer Masked Assessment
Description: At least 2 out of 3 blinded Independent Photographic Reviewers (IPRs) correctly identify the 90-day image of a subject from the pair of baseline and 90-day images.
Time Frame: 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants | 55

3. Other Pre Specified Outcome: Investigator Fitzpatrick Wrinkle and Elastosis Scale
Description: Magnitude of improvement measured by the mean change in FWS from baseline, 90-day, 180-day visit as determined by Investigators. Scale ranges from 1 (no wrinkles) to 9 (most wrinkles).
Time Frame: Baseline, 90-day Change, 180-day Change
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
score on a scale
  Baseline | 7.4 (1.1)
  90 Day Change | -4.4 (1.8)
  180 Day Change | -4.4 (2.0)

4. Other Pre Specified Outcome: Subject Global Aesthetic Improvement Scale
Description: Subject rated GAIS: Very much improved, much improved, improved, no change, worse, much worse, very much worse
Time Frame: 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants
  Very Much Improved | 27
  Much Improved | 21
  Improved | 5
  No Change | 2
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

5. Other Pre Specified Outcome: Investigator Global Aesthetic Improvement Scale
Description: Investigator rated GAIS: Very much improved, much improved, improved, no change, worse, much worse, very much worse
Time Frame: 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants
  Very Much Improved | 36
  Much Improved | 17
  Improved | 2
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

6. Other Pre Specified Outcome: Patient Satisfaction Questionnaire
Description: 5 questions pertaining to satisfaction with results, would you recommend to a friend, would you have the procedure done again, any changes noticed, and any improvement in quality of life.
Time Frame: 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants
  Happy With Results of Procedure | 53
  Would Recommend Procedure to a Friend | 46
  Would Consider Having the Procedure Performed Again | 35
  Which Changes do You See in the Area Treated: None | 0
  Skin Texture Improvement | 52
  Skin Tone Improvement | 47
  Skin Pigmentation Improvement | 36
  Fine Lines and Wrinkles Improvement | 50
  Skin Pore Size Improvement | 40
  Skin Feels Better | 44
  Skin Feels Tighter | 51
  Skin Looks Tighter | 52
  Skin Looks More Radiant | 41
  Skin Appears Brighter | 38
  Skin Seems More Youthful | 50
  Other Changes Noted | 6

7. Other Pre Specified Outcome: Pain and Discomfort
Description: Evaluation of the change in pain and discomfort after treatment (baseline, within 60 minutes following the procedure) as reported by the subject on a visual analog scale (VAS)experienced in the period up to the 10-day follow-up visit. Any pain or discomfort will be recorded daily by each participant in a diary using an 11-point Visual Analogue Scale (VAS) where 0 is no pain and 10 is most pain.
Time Frame: Baseline to Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
score on a scale
  Baseline | 0.0 (0.0)
  Post-Procedure | 3.7 (2.8)
  1 Day | 2.4 (2.6)
  6 Day | 2.9 (2.6)
  10 Day | 1.1 (1.6)

8. Other Pre Specified Outcome: Percentage of Subjects With Achievement of Re-Epithelialization
Description: Achievement of re-epithelialization by facial zone and across all facial zones as reported by the investigator.
Time Frame: 10-day, 30-day, 90-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants
  10 Day | 3
  30 Day | 48
  90 Day | 55

9. Other Pre Specified Outcome: Comfortable in Public
Description: Mean duration until study subject feels comfortable going in public after treatment as reported by the study subject. Willing to go out in public by the 10-day visit.
Time Frame: 10-day
Measure: Count of Participants; unit: Participants
Arm/Group | Full-face Renuvion Dermal System Treatment
Number analyzed (Participants) | 55
Participants | 28

ADVERSE EVENTS:
Time Frame: Through 6 month follow-up visit for all enrolled subjects.
Arm/Group | Full-face Renuvion Dermal System Treatment
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 1/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full-face Renuvion Dermal System Treatment (N=55)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — The subject was admitted to the hospital for bowel obstruction. After Investigator review, this event was identified to be secondary to prior bowel cancer that was not reported by subject at baseline. This is not related to study device or procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full-face Renuvion Dermal System Treatment (N=55)
Erythema/skin inflammation/ focal skin congestion (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 55 (56)
Crusting (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 55 (55)
Edema/Swelling (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 55 (55)
Pain/Tenderness (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 30 (30)
Milia/acne (Skin and subcutaneous tissue disorders) | 16 (20)
Pruritus/itching (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 14 (14)
Hypertrophic scarring (Skin and subcutaneous tissue disorders) | 8 (8)
Post-inflammatory hyperpigmentation (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 6 (6)
Telangiectasias (Skin and subcutaneous tissue disorders) | 6 (6)
Discoloration/hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Pinpoint Bleeding (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 2 (2)
Prolonged Wound Healing (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria/rash (Expected Treatment Effect) (Skin and subcutaneous tissue disorders) | 2 (2)
Eye Irritation (Eye disorders) | 1 (1)
Nausea during Procedure (Gastrointestinal disorders) | 3 (3)
Emesis/Vomiting Post-Procedure (Gastrointestinal disorders) | 2 (2)
Drug Reaction During Procedure (General disorders) | 1 (1)
Lower Lid Retraction (Eye disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — Unrelated to device/procedure
Self-Inflicted Superficial Excoriations (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study include the lack of an ideal internal control as is typically the case in facial skin resurfacing studies and in single-arm studies, inability to precisely control energy density across study sites and between subjects, inability to ensure uniformity of aftercare measures employed by subjects as well as limited post-treatment follow-up of just 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04185909/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04185909/SAP_001.pdf